CLINICAL TRIAL: NCT06370247
Title: First-time Usage of SGLT2 Inhibitors in Type 2 Diabetic Patients Who Are Fasting During Ramadan: Safety and Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Ahmed Mohamed, lecturer of internal medicine, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-04-07PD.
Record Dates: First submitted 2023-11-07; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: SGLT2 Inhibitors, First Time Use; Type2 Diabetes; Fasting in Ramadan
Keywords: SGLT2 inhibitors; type 2 DM; fasting inramadan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients With T2DM, willing to fast Ramadan and treated with SGLT2 inhibitors (Other): Egyptian male and female Muslim patients, aged ≥ 18 years old. With T2DM, willing to fast Ramadan and treated with SGLT2 inhibitors (empagliflozin, dapagliflozin) as an add-on to metformin or other oral hypoglycemic agent.
  Interventions: Diagnostic Test: HbA1c, serum creatinine, eGFR urine analysis and serum electrolyte Na and K

INTERVENTIONS:
Diagnostic Test: HbA1c, serum creatinine, eGFR urine analysis and serum electrolyte Na and K — HbA1c, serum creatinine, eGFR urine analysis and serum electrolyte Na and K will measure

SUMMARY:
All healthy Muslim adults are required to observe the Ramadan fast, which is one of Islam's five pillars. People with Type 2 Diabetes Mellitus frequently fast throughout Ramadan (T2DM).

Although fasting during Ramadan is said to have positive effects on diabetes patients, such as a reduction in excess body weight and an improvement in lipid profile it can be linked to a slight increased risk for metabolic complications that need immediate attention, such as hypoglycemia and hyperglycemia, dehydration, and diabetic ketoacidosis (DKA The number of diabetics worldwide was projected to reach 537 million in 2021. Studies have shown that there are a rising number of people in this category, and by 2045, there will be 738 million people worldwide who have diabetes. Almost 150 million Muslims worldwide have diabetes, and this number is progressively rising. Research estimates that 118 million of these Muslims who have diabetes fast throughout Ramadan, underscoring the need of choosing the best treatment strategy at this time. Almost two-thirds of all Muslims with T2DMfast throughout the month of Ramadan, according to studies from CREED, Epidemiology of Diabetes, and Ramadan.According to this, the most recent study showed that 86% of patients with T2DMreported a fast for at least 2 weeks.

Patient education, which should cover information on risks, lifestyle modifications, glucose monitoring, diet, exercise, and medication, is a crucial component of managing diabetes during Ramadan.Several studies have demonstrated the effectiveness and safety of sodium glucose cotransporter 2 inhibitors (SGLT2 I) in T2DM patients who are fasting throughout Ramadan. In individuals with T2DM, SGLT2 inhibitors have shown to reduce cardiovascular events and slow the course of renal disease.

In the literature published so far, SGLT2i has shown lower rates of hypoglycemia and hypovolemia during fasting as compared to sulphonylureas (SU).

ELIGIBILITY:
Inclusion Criteria:

* Egyptian male and female Muslim patients,
* aged ≥ 18 years old.
* patients with T2DM
* willing to fast Ramadan and treated with SGLT2 inhibitors (empagliflozin, dapagliflozin) as an add-on to metformin or other oral hypoglycemic agent.

Exclusion Criteria:

* *Patients with chronic liver disease (serum levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase above 2 times upper limit of normal value).

  * Patients with chronic renal disease (estimated glomerular filtration rate (eGFR) <25 ml/min/1.73 m2).
  * Patients on renal dialysis
  * patients with a history of ketoacidosis in the past six months patients had a history of malignancy during the past three years.
  * Also, subjects with strokes including transient ischemic attack (TIA),
  * patients with diabetic foot infection, amputation (non-traumatic even minor), or gangrene were excluded.
  * In addition to pregnant or breast-feeding women.
  * Besides, those who had a history of frequent urinary tract infections (UTI) were also excluded from the study.

Patients who will discontinue the SGLT2i during Ramadan and those who will fast for less than 15 days will be excluded from the final analysis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
blood glucose level monitoring | 6 weeks after ramadan
  measurement of HbA1c in percent
safety of SGLT2 inhibitors usage during ramadan | 6 weeks after ramadan
  measurement of serum creatinine mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khalil HAM, Abdelal SK, El-Rawy AF, Abodahab ALH. First-Time Usage of SGLT2 Inhibitors in Patients With Type 2 Diabetes Who Are Fasting Ramadan: Efficacy and Safety. J Diabetes Res. 2025 Apr 25;2025:4321423. doi: 10.1155/jdr/4321423. eCollection 2025. PMID 40322737